CLINICAL TRIAL: NCT07108634
Title: Cost-effectiveness Analyses for the Prevention of Acute Kidney Injury in Patients Undergoing Cardiac Surgery in the UK
Acronym: Cost-AKI
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025CAR140
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
Keywords: Cardiac surgery; Cardiopulmonary bypass machine
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who developed AKI in their post-operative phase: Consecutive patients who have undergone cardiac surgery at the various cardiac surgery centres in the UK and who developed AKI in their post-operative phase will be selected.
  Interventions: Other: RenalGuard Therapy
- Patients who did not develop AKI in their post-operative phase: The patients who developed AKI group will be propensity-matched 1:1 to patients who did not develop AKI

INTERVENTIONS:
Other: RenalGuard Therapy — The RenalGuard Therapy® is comprised of a console, a single-use sterile IV infusion set, urine collection set and a cart. The console is a microcontroller device that has a means for measuring urine output and automatically controls the hydration infusion pump based on the measured urine output and clinician settings. The system is designed for infusion of hydration solutions only. The patient is connected to the console by the IV Infusion set connected to the patient's peripheral IV cannula and the urine collection set connected to the patient's indwelling Foley urinary catheter. The console continuously monitors urine production by measuring the weight of urine in the collection set, converts the urine weight to volume and then, automatically infuses the pre-set volume of hydration fluid to compensate for this output.
  Groups: Patients who developed AKI in their post-operative phase

SUMMARY:
Multi-centre retrospective analysis of prospectively collected data with propensity matched scoring groups (AKI v/s non-AKI). Data collection from databases (or their equivalent): PATS Dendrite, Electronic Medical Records, TD-web (results Portal), MedTrack (ICU database), iSite (Radiology), SPY (Long-term status)

DETAILED DESCRIPTION:
1.1 BACKGROUND Cardiac surgery associated acute kidney injury (CSA-AKI) is reported in 25-40% of patients. This variability is due to a spectrum of definitions used to classify AKI. AKI definition and staging are based on the Risk, Injury, Failure, Loss, End-stage kidney disease (RIFLE) criteria and the Acute Kidney Injury Network (AKIN) criteria, which have been further refined in the Kidney Disease: Improving Global Outcomes (KDIGO) AKI work group guidelines. It is now customary to use the KDIGO definition or its modified version - the AKIN consensus criteria. The development of AKI in the post-op cardiac surgery setting is associated with significant morbidity, mortality, prolonged intensive care (ICU) & in-hospital stays, increased treatment costs and poorer long-term survival and quality of life. Till now, no satisfactory strategy has been successful in preventing CSA-AKI despite the pre-operative knowledge of those patients who are at risk of developing it.

RenalGuard Therapy® (Cardiorenal Systems, Boston, USA) is an automated fluid management system which measures the volume of urine output and enables the physician to set a personalized, instantaneous fluid replacement rate based on the measured urine output. The RenalGuard Therapy® is comprised of a console, a single-use sterile IV infusion set, urine collection set and a cart. The console is a microcontroller device that has a means for measuring urine output and automatically controls the hydration infusion pump based on the measured urine output and clinician settings. The system is designed for infusion of hydration solutions only. The patient is connected to the console by the IV Infusion set connected to the patient's peripheral IV cannula and the urine collection set connected to the patient's indwelling Foley urinary catheter. The console continuously monitors urine production by measuring the weight of urine in the collection set, converts the urine weight to volume and then, automatically infuses the pre-set volume of hydration fluid to compensate for this output. The system is placed on a cart that is designed to hold the console, infusion set, and urine collection set. Safety mechanisms and patient's protection have been designed and incorporated into the RenalGuard Therapy® to support appropriate balance and rates of IV infusion without fluid overloading or dehydrating the patient.

The use of the RenalGuard® Therapy was initially investigated at reducing AKI in patients at risk of contrast-induced nephropathy (CIN) when undergoing either percutaneous coronary intervention (PCI) or transcatheter aortic valve implantation (TAVI). These studies showed that in patients with chronic kidney disease, the RenalGuard® Therapy reduced the incidence of AKI by 60 to 75% as compared to controls.

The use of the RenalGuard® Therapy in patients undergoing cardiac surgery has only been reported recently. The recent RCT data showed that in patients at risk of developing AKI during cardiac surgery, the RenalGuard® Therapy reduced CSA-AKI rate from 20.9% to 10%.

1.2 RATIONALE FOR CURRENT STUDY AKI is known to be associated with significant costs in healthcare delivery in patients undergoing cardiac surgery. It is estimated that AKI in that group of patients could increase costs by $19,212. In a more recent study published in 2018, the estimated additional cost for AKI post cardiac surgery was reported at $38,358 with a 10-fold increase in mortality (13.9% vs 1.3%) as well as a doubling in the in-hospital stay (mean 18.2 vs 8.6 days) when compared to non-AKI patients. ICU stay has also been reported to be prolonged in patients, post CABG, who developed AKI (mean 5.5 vs 2.2 days).

The KIDNEY study confirmed the clinical benefit for the RenalGuard® Therapy. However, the RenalGuard® Therapy does come at a cost and no cost-effectiveness data is currently available in the literature. It is important within the UK NHS setting to assess whether this clinical benefit to the patient has also some cost-effectiveness value attached to it, given that RenalGuard Therapy is marketed at €1,000 per patient in Europe.

2. STUDY OBJECTIVES Primary objective: Cost-effectiveness assessments using QALY gained & ICER, with the use of the RenalGuard® Therapy for the reduction of CSA-AKI in patients undergoing cardiac surgery.

Secondary objectives: CSA-AKI incidence (as defined by modified KDIGO), ICU & in-hospital stays, costs of ICU and in-hospital stays and survival rates (index admission and follow-up at the time of the study), best cost-effectiveness sub-group(s).

3. STUDY DESIGN This is a multi-centre, propensity-matched, retrospective study involving patients who developed AKI after cardiac surgery (CSA-AKI) compared to 1:1 propensity-matched scoring non-AKI patients.

It involves retrieving patient's clinical data which was prospectively recorded during the patients stay when they underwent cardiac surgery at various cardiac surgery centres in the UK. The data are currently within the PATS Dendrite, Electronic Medical Records, TD-web (results Portal), MedTrack (ICU database), iSite (Radiology), SPY (Long-term status) databases, or their equivalents.

The PATS dendrite database records pre-op, intra-op and post-op data pertaining to patient characteristics, operative details, ICU and ward stay including complications. Data recorded include date of operation, patient's age, body mass index & gender, risks factors (diabetes, left ventricular function, urgency of procedure), type of procedure, Log Euroscore, cardiopulmonary bypass time, date of extubation, need for inotropes, any complications (respiratory including additional respiratory support, re-exploration, arrhythmias, neurological dysfunction, renal dysfunction, blood transfusion, gastro-intestinal problems), date of ICU discharge, ICU re-admission, date of hospital discharge, patient status at time of discharge and discharge destination. This data is independently verified by the cardiac audit personnel and then the core data is submitted to NICOR from where surgeon-specific and Unit-specific mortality data is confirmed and published on the DoH/SCTS website.

The MedTrack Database records the patient's complications and length of stay on the ICU.

The iSite details all the radiological investigations while the TD-Web includes all the investigations results (e.g. blood analysis). Data on all databases are recorded contemporaneously. The Clinical Web Portal (Electronic Medical Records) will be used to cross check this information. Some data may need to be retrieved from the medical records.

Survival data will be retrieved from the SPY database while hospital cost data will be requested from the hospital finance department.

This study (data collection) will run over a period of six months. Thereafter, data analysis & interpretation, manuscript writing & publication may take up to another six months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiac surgery (elective or in-house urgent) from Jan 1st, 2013, to December 31st, 2023 (excluding patients during 2020 & 2021 - due to confounding Covid-19 impact on AKI)
2. Cardiopulmonary bypass machine was used during cardiac surgery
3. Patient's data available in the databases (Minimum dataset required for propensity matching: age, gender, diabetes history, LVEF, priority of surgery, pre-op haemoglobin & SCr levels, cardiac surgery performed, CPB duration, Euroscore or LogEuroscore, RRT use, post-op D1&/or D2 &/or D3 SCr)

Exclusion Criteria:

1. Emergency surgery
2. Patient with incomplete dataset*
3. Surgery performed without CPB
4. Patients already dialysis dependent
5. Patient with eGFR <20 mL/min/1.73 m²
6. Cardiac surgery requiring deep hypothermic circulatory arrest (DHCA)
7. Patients previously treated with RenalGuard® Therapy
8. Patient has opted-out of research (data opt-out) * Data completeness - These variables need to be complete for the propensity matching: age, gender, diabetes history, LVEF, priority of surgery, pre-op haemoglobin & SCr levels, cardiac surgery performed, CPB duration, Euroscore or LogEuroscore, RRT use, post-op D1&/or D2 &/or D3 SCr

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who have undergone cardiac surgery at the various cardiac surgery centres in the UK and who developed AKI in their post-operative phase will be selected. This group will be propensity-matched 1:1 to patients who did not develop AKI. A total of around 8000 patients' data will be accessed to obtain approximately 4000 patients' (2,000 in each group) data for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
CSA-AKI | 6 months
  If there is an increase in serum creatinine (SCr) by ≥0.3 mg/dl (≥26.5 micromol/l) within 72 hours of surgery compared to the baseline value
CSA-AKI | 6 months
  If there is an increase in SCr by ≥1.5 times from SCr value at baseline within 72 hours of surgery; or use of RRT within 7 days of surgery.

SECONDARY OUTCOMES:
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  CSA-AKI incidence
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  ICU stay duration
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  In-hospital stay duration
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  In-hospital survival
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  Survival at time of study
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  Costs of ICU stay (HRG)
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  Costs of in-hospital stay
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  Cost benefit & cost effectiveness calculations if CSA-AKI were to be reduced using the RenalGuard® Therapy: QALY gained, ICER
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  If cost benefit applies to all patient groups or to specific patient group (sub-group analysis e.g. CKD, Diabetes, elderly - over 70 years)
CSA-AKI patient group vs non CSA-AKI patient group | 6 months
  Cost of RenalGuard® Therapy at which it is no longer cost-effective.

CONTACTS AND LOCATIONS:
Locations (1):
- New Cross Hospital, Wolverhampton, West Midlands, United Kingdom